CLINICAL TRIAL: NCT04083612
Title: Evaluation of the Predictive Value of Early Serum Trough Concentrations and Anti-drug Antibodies of Ixekizumab and the Development of Concentration-response Curve of Ixekizumab for Psoriasis Patients
Brief Title: Therapeutic Drug Monitoring of Ixekizumab in Psoriasis Patients
Acronym: BIOLOPTIM-IXE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: KU Leuven (Other); University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-05355 - BIOLOPTIM-IXE
Record Dates: First submitted 2019-07-19; First posted 2019-09-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Psoriasis Vulgaris
Keywords: Psoriasis; Therapeutic drug monitoring; Ixekizumab
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: A prospective, open label, non-randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standard of care - ixekizumab (Other): Patient will continue to receive ixekizumab according to standard of care dosing regimen, i.e. loading dose first (160 mg) at week 0; 80 mg every 2 weeks until week 12, then 80 mg every 4 weeks
  Interventions: Procedure: Venapuncture; Other: Patient questionnaires

INTERVENTIONS:
Procedure: Venapuncture — Blood samples will be collected to determine the serum trough levels and anti-drug antibodies of ixekizumab
Other: Patient questionnaires — The study participant will complete the Dermatology Quality of Life Index (DLQI) and EQ5D5L questionnaires at each study visit.

SUMMARY:
Biologics, such as ixekizumab, are currently the most effective treatment option for patients with moderate-to-severe psoriasis. But they are costly for health care systems and prescribed according to a 'one dose fits all' dosing regimen, leading to potential over- and undertreatment. Within this study the investigators aim to investigate the predictive value of early serum trough levels of ixekizumab and determine the therapeutic window of ixekizumab in psoriasis patients.

DETAILED DESCRIPTION:
Patients will be included after siging informed consent. After inclusion, patients will continue on standard dosing schedule of ixekizumab (i.e. one loading dose of 2 subcutaneous injections (160 mg) at week 0, followed by one subcutaneous injection (80 mg) every 2 weeks for 12 weeks, and then one subcutaneous injections (80 mg) every 4 weeks). During each study visit, blood will be taken in order to quantify Ctroughs and/or anti-drug antibodies towards ixekizumab. In addition, the Psoriasis Severity and Area Index (PASI) and the Investigator's Global Assessment (IGA) score will be evaluated by a physician. Patients complete the Dermatology Life Quality Index (DLQI) and European quality of life EQ-5D instrument at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have a clinical or histological diagnosis of chronic plaque-type psoriasis
2. Participants must sign an ICF indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study

Exclusion Criteria:

1. Participants who have currently a predominant nonplaque form of psoriasis
2. Participants who are pregnant, nursing or planning a pregnancy
3. Participants who are unable or unwilling to undergo multiple venapunctures
4. Participants who are treated according to a different dosing schedule than standard dosing of ixekizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Predictive value of early serum trough concentrations of ixekizumab | Week 0 until week 24 of treatment
  Prediction of the clinical response (PASI) at week 12 and/or week 24 based on serum trough concentrations measurements taken from week 0, 1, 2, 3 and/or 4.
Predictive value of early anti-drug antibodies of ixekizumab | Week 0 until week 24 of treatment
  Prediction of the clinical response (PASI) at week 12 and/or week 24 based on anti-drug antibodies measurements taken from week 0, 1, 2, 3 and/or 4.
The development of a therapeutic window of ixekizumab in psoriasis | Week 0 until week 52 of treatment
  Defining a therapeutic window for ixekizumab based on serum trough levels corresponding with adequate clinical response.

SECONDARY OUTCOMES:
DLQI | Week 0 until week 52 of treatment
  The DLQI (Dermatology Life Quality Index) (range 0-30) is a dermatology specific quality of life (QoL) instrument designed to assess the impact of the disease on participant's QoL. It is a ten item questionnaire that, in addition to evaluated overall QoL, can be used to assess six different aspects that may affect QoL: 1) symptoms and feelings, 2) daily activities, 3) leasure, 4) work or school performances, 5) personal relationships, and 6) treatment.
  The scoring of each question is as follows:
  Very much - scored 3; A lot - scored 2; A little - scored 1; Not at all - scored 0; Not relevant - scored 0; Question 7, 'prevented work or studying' - scored 3. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
EQ5D5L | Week 0 until week 52 of treatment
  The 5-level EQ-5D version (EQ-5D-5L) was introduced by the EuroQol Group in 2009 to improve the instrument's sensitivity and to reduce ceiling effects.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems (level 1), slight problems (level 2), moderate problems (level 3), severe problems (level 4) and extreme problems (level 5). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state, which is the outcome result. There is no minimum or maximum score since the the 5 digit-number is a non-numeric variable.
EQ VAS | Week 0 until week 52 of treatment
  The EQ VAS (Visual Analogue Scale) (range 0-10) records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement. Minimum score is 0%, max. score is 100%. Lower values mean 'worse health the patient can imagine', higher values mean 'better health the patient can imagine'.

CONTACTS AND LOCATIONS:
Overall Officials: Jo Lambert, Prof., Principal Investigator — University Ghent
Locations (7):
- Belgium (7):
  - AZ Maria Middelares, Ghent, Oost-Vlaanderen
  - AZ Sint-Lucas, Ghent, Oost-Vlaanderen
  - University Hospital of Ghent, Ghent, Oost-Vlaanderen
  - Private Practice Dermatology, Maldegem, Oost-Vlaanderen
  - UZ Hospital, Leuven, Vlaams-Brabant
  - AZ Sint-Jan, Bruges, West-Vlaanderen
  - AZ Delta Rembert, Torhout, West-Vlaanderen

IPD SHARING:
Plan to Share IPD: No